CLINICAL TRIAL: NCT07025174
Title: Evaluation of the Effect of Sequential Anti-angiogenic Therapy Following Immune Therapy Progression on Survival in Patients With Advanced Biliary Tract Malignancies: A Randomized, Multi-center, Exploratory Clinical Study
Brief Title: Sequential Anti-Angiogenic Therapy After Immunotherapy in Advanced Biliary Tract Cancer
Acronym: SAIB
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT20250065C-R1
Record Dates: First submitted 2025-06-10; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: Bile Duct Carcinoma; Gall Bladder Cancer; Biliary Tract Cancer; Cholangiocarcinoma
Keywords: Biliary tract cancer; Immunotherapy; Anti-angiogenic therapy; Anlotinib; Sequential therapy
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms; Biliary Tract Neoplasms; Cholangiocarcinoma | interventions — Gemcitabine; Cisplatin; anlotinib; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Chemotherapy First-line (Active Comparator): Patients receive standard gemcitabine plus cisplatin (GP) chemotherapy as first-line treatment for up to 6 cycles. Upon disease progression, patients receive second-line treatment with XELOX or FOLFOX chemotherapy plus anlotinib.
  Interventions: Drug: Gemcitabine, Cisplatin; Drug: Anlotinib; Drug: Oxaliplatin + 5-Fluorouracil/Leucovorin
- Immunotherapy Plus Chemotherapy First-line (Experimental): Patients receive gemcitabine plus cisplatin (GP) chemotherapy combined with PD-1/CTLA-4 dual functional antibody as first-line treatment for up to 6 cycles. Upon disease progression, patients receive the same second-line treatment as the control group with XELOX or FOLFOX chemotherapy plus anlotinib.
  Interventions: Drug: PD-1/CTLA-4 Dual Functional Antibody; Drug: Gemcitabine, Cisplatin; Drug: Anlotinib; Drug: Oxaliplatin + 5-Fluorouracil/Leucovorin

INTERVENTIONS:
Drug: PD-1/CTLA-4 Dual Functional Antibody — PD-1/CTLA-4 Dual Functional Antibody (iparomlimab and tuvonralimab injection):
  5 mg/kg intravenous infusion every 3 weeks (day 1 of each 21-day cycle) for up to 6 cycles, with potential for maintenance therapy continuation. Used in combination with GP regimen in experimental arm only. This is a novel dual-functional antibody targeting both PD-1 and CTLA-4 pathways simultaneously.
  Arms: Immunotherapy Plus Chemotherapy First-line
Drug: Gemcitabine, Cisplatin — Gemcitabine 1000 mg/m² d1,8+Cisplatin 25mg/m² d1,8
Drug: Anlotinib — 10mg po d1-14 q3w
Drug: Oxaliplatin + 5-Fluorouracil/Leucovorin — XELOX (oxaliplatin 130mg/m² d1+capecitabine 1000mg/m² d1-14 q3w) or FOLFOX6 (Oxaliplatin 85 mg/m², leucovorin 400 mg/m², fluorouracil 400 mg/m² intravenous bolus followed by fluorouracil 2400 mg/m² 46 hours, q2w)

SUMMARY:
Brief Summary:

This study is for patients with advanced biliary tract cancer (cancer of the bile ducts or gallbladder). The purpose is to find out if using anti-blood vessel formation drugs after immunotherapy treatment can help patients live longer without their cancer getting worse.

What the study compares:

Control group: Patients receive standard chemotherapy as first-line treatment, then chemotherapy plus anlotinib (an anti-blood vessel drug) if their cancer progresses Treatment group: Patients receive chemotherapy plus immunotherapy as first-line treatment, then the same second-line treatment as the control group if their cancer progresses

Who can join:

Patients aged 18-75 with advanced biliary tract cancer that has been confirmed by tissue testing, who have not received immunotherapy or anti-blood vessel drugs before, and who are in good enough health for treatment.

What we want to learn:

The main goal is to see if patients who received immunotherapy first have better outcomes when they later receive anti-blood vessel treatment. We will measure how long patients live without their cancer getting worse during second-line treatment.

Study design:

This is a randomized study, meaning patients are assigned by chance to one of the two treatment groups. About 60 patients will participate across multiple hospitals in China. We will also collect blood and tissue samples to better understand how these treatments work.

The study will help doctors determine if this treatment sequence could become a new standard approach for patients with advanced biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

Age 18-75 years at time of enrollment; Histologically or cytologically confirmed advanced or metastatic biliary tract adenocarcinoma (intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, or gallbladder carcinoma); Unresectable locally advanced or metastatic disease not amenable to curative treatment; At least one measurable lesion according to RECIST version 1.1 criteria; ECOG Performance Status 0-1; Life expectancy ≥ 12 weeks; No prior systemic chemotherapy, immunotherapy, or anti-angiogenic therapy for advanced disease (adjuvant therapy completed >6 months prior is allowed); Adequate bone marrow function: ANC ≥1.5×10⁹/L, platelets ≥100×10⁹/L, hemoglobin ≥90 g/L; Adequate liver function: Total bilirubin ≤2.5×ULN, ALT and AST ≤3×ULN (or ≤5×ULN if liver metastases present); Adequate renal function: Serum creatinine ≤1.5×ULN or creatinine clearance ≥50 mL/min; Signed informed consent.

Exclusion Criteria:

Mixed histology tumors or neuroendocrine components; Active central nervous system metastases (treated and stable metastases >4 weeks allowed); History of other malignancies within 5 years (except adequately treated basal cell carcinoma, squamous cell carcinoma of skin, or carcinoma in situ); Active autoimmune disease requiring systemic treatment; History of severe allergic reactions to monoclonal antibodies or study drug components; Uncontrolled hypertension (>140/90 mmHg despite medication); Significant cardiovascular disease including unstable angina, myocardial infarction within 6 months, or NYHA Class III-IV heart failure; Active bleeding or bleeding tendency, thrombosis, or use of anticoagulants; Major surgery within 4 weeks or minor surgery within 2 weeks; Active infection requiring systemic treatment; Pregnancy or breastfeeding; HIV infection, active hepatitis B or C infection; Psychiatric illness that would limit compliance with study requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) of Second-Line Treatment | From the start of second-line treatment until disease progression or death from any cause, assessed up to 24 months
  Progression-free survival defined as the time from initiation of second-line chemotherapy plus anlotinib treatment until radiographic disease progression per RECIST 1.1 criteria or death from any cause, whichever occurs first. Disease progression will be assessed by CT or MRI imaging every 2 treatment cycles (approximately every 6 weeks). This outcome measure specifically evaluates whether patients who received first-line immunotherapy plus chemotherapy have improved PFS during second-line anti-angiogenic treatment compared to patients who received first-line chemotherapy alone.

CONTACTS AND LOCATIONS:
Overall Officials: Tingbo Liang, MD, Principal Investigator — Department of Hepatobiliary and Pancreatic Surgery, The First Affiliated Hospital, Zhejiang University School of Medicine
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided